CLINICAL TRIAL: NCT04015232
Title: An Assessor-blind, Balanced, Parallel, Randomized, Two-treatment, Comparative Immunogenicity Study of Multiple Doses of INTP5 of Intas Pharmaceuticals Limited, India Against Neulasta® of Amgen Inc., USA Administered Subcutaneously in Healthy, Adult, Human Subjects Under Fed Condition.
Brief Title: Comparative Immunogenicity Study of Multiple Doses of Proposed Pegfilgrastim Biosimilar, INTP5 of Intas Pharmaceuticals Ltd., India Against Neulasta of Amgen Inc., USA in Healthy, Adult Human Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intas Pharmaceuticals, Ltd. (Industry)
Collaborators: Lambda Therapeutic Research Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0554-17
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Immunogenicity; Healthy Volunteers
Keywords: Pegfilgrastim; Biosimilar; Immunogenicity; Pharmacokinetics; Pharmacodynamics; Safety; Healthy Volunteers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study staff taking care of subject's safety and the laboratory personnel doing the sample analysis of PK, PD, and immunogenicity data were blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- INTP5 biosimilar product (Experimental): INTP5 subcutaneously at a dose of 6 mg/0.6 mL.
  Interventions: Combination Product: INTP5
- US Neulasta reference product (Active Comparator): US Neulasta subcutaneously at a dose of 6 mg/0.6 mL.
  Interventions: Combination Product: US Neulasta

INTERVENTIONS:
Combination Product: INTP5 — INTP5, a pegfilgrastim biosimilar to US Neulasta.
  Arms: INTP5 biosimilar product
Combination Product: US Neulasta — US Neulasta: FDA approved pegfilgrastim innovator product.
  Arms: US Neulasta reference product

SUMMARY:
The study was an assessor-blind, balanced, parallel, randomized, two-treatment, comparative immunogenicity study of multiple doses of subcutaneous (SC) Pegfilgrastim injection (6 mg/0.6 mL; Intas Pharmaceuticals Ltd. proposed biosimilar INTP5 compared to innovator product, US-Neulasta) in healthy, adult, human subjects under fed conditions.

ELIGIBILITY:
Inclusion criteria:

1. Normal, healthy adult human volunteers between 18 to 45 years of age (both inclusive) living in and around Ahmedabad city or western part of India.
2. Having body weight ≥50 kg and body mass index (BMI) between 18.5 and 29.9 (both inclusive), calculated as weight in kg/height in meter^2.
3. Not having any significant disease in medical history or clinically significant abnormal findings during screening, abdominal ultrasonography, medical history, clinical examination, laboratory evaluations, 12-lead echocardiogram (ECG) and chest X-ray (posterior-anterior view; within the last 6 months) recordings.
4. Able to understand and comply with the study procedures, in the opinion of the investigator.
5. Able to give voluntary written informed consent for participation in the trial.
6. In case of female subjects:

   * Surgically sterilized at least 6 months prior to study participation; Or If a woman of child bearing potential is willing to use a suitable and effective double barrier contraceptive method or intra uterine device during the study.
   * Serum pregnancy test (for female subjects) must be negative.

Exclusion criteria:

1. Known hypersensitivity to the study drug or its constituents and/or hypersensitivity to E. coli derived proteins, and/or previous exposure to the study drug.
2. History or presence of any disease or condition which might compromise the haemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system.
3. Known case of hereditary fructose intolerance.
4. Subjects with latex allergies will be excluded as the needle cover on the single-use prefilled syringe contains dry natural rubber (latex).
5. Any clinically significant laboratory finding including absolute neutrophil count (ANC), platelet, red blood cells (RBC) count, and hemoglobin level at the time of screening.
6. Prior exposure to any peptide colony stimulating or growth factor, including erythropoietin, filgrastim or Pegfilgrastim; Prior exposure to any vaccines, immunoglobulin preparations or immunomodulators within the past 6 months prior to receiving first dose; evidence of E. coli diarrhea or diseases within 3 months.
7. Any history or presence of asthma (including aspirin-induced asthma) or nasal polyp or NSAIDs induced urticaria.
8. Subjects with a history of pulmonary infiltrate or pneumonia in the last 6 months.
9. History of any hematologic disease including sickle cell disorders.
10. Ingestion or use of any prescribed medication at any time within 1 month prior to receiving first dose.
11. Receipt of over-the-counter medicines which have not yet cleared from the body (5 half-lives must have passed for the medicine to be considered to have cleared from the body).
12. A recent history of harmful use of alcohol, i.e. alcohol consumption of more than 14 standard drinks per week for men and more than 7 standard drinks per week for women (A standard drink is defined as 360 mL of beer or 150 mL of wine or 45 mL of 40% distilled spirits, such as rum, whisky, brandy etc.) or consumption of alcohol or alcoholic products within 72 hours prior to receiving study medicine.
13. Smokers, who smoke 10 or more than 10 cigarettes/day or inability to abstain from smoking during the study.
14. Use of any recreational drugs or history of drug addiction or testing positive in pre-study drug scans.
15. Donation of blood (1 unit or 350 mL) or equivalent amount of blood substitute.
16. Receipt of an investigational medicinal product or participation in a drug research study within a period of 90 days prior to the first dose of study medication. Elimination half-life of the study drug should be taken into consideration for inclusion of the subject in the study.
17. Positive result for human immunodeficiency virus (HIV I &/or II) and/or hepatitis B and C tests.
18. History or presence of cancer because of which anticipated life span is less than 5 years as per the investigator's assessment.
19. History or presence of psychiatric disorders.
20. Presence of tattoo or scars or any type of skin lesions due to infection, burning, wound or inflammation at the proposed site of injection.
21. An unusual diet, for whatever reason (e.g. low-sodium), for 4 weeks prior to receiving the study medicine. In any such case, subject selection will be at the discretion of the Principal Investigator.
22. Consumption of grape fruit or grape fruit products within 72 hours prior to receiving study drug.
23. A history of difficulty in donating blood.
24. Females, pregnant or lactating, or planning to become pregnant during the time the subject is on study or found positive in pregnancy test at screening.
25. Any infections in the last 4 weeks before receiving study medication.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adarsh K Garg, M.B.B.S, Principal Investigator — Lambda Therapeutic Research Ltd.; Vinu Jose, M.D., Study Director — Intas Pharmaceuticals, Ltd.
Locations (1):
- Lambda Therapeutic Research Ltd., Ahmedabad, Gota, India

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- INTP5 Biosimilar Product: INTP5 subcutaneously at a dose of 6 mg/0.6 mL.
  INTP5: A pegfilgrastim biosimilar to US Neulasta.
- US Neulasta Reference Product: US Neulasta subcutaneously at a dose of 6 mg/0.6 mL.
  US Neulasta: FDA approved pegfilgrastim innovator product.
Period: Overall Study
Arm/Group | INTP5 Biosimilar Product | US Neulasta Reference Product
Started | 100 | 100
Completed | 89 | 93
Not Completed | 11 | 7
Not completed — Withdrawal by Subject | 7 | 4
Not completed — Protocol Violation | 1 | 0
Not completed — Medical Grounds | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | INTP5 Biosimilar Product | US Neulasta Reference Product | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (6.82) | 34.3 (6.05) | 32.9 (6.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 60 | 60 | 120
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 100 | 100 | 200
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  India | 100 | 100 | 200
Height [Mean (Standard Deviation); unit: cm] | 160.2 (8.48) | 160.1 (8.68) | 160.2 (8.56)
Weight [Mean (Standard Deviation); unit: kg] | 61.3 (8.31) | 62.6 (7.49) | 61.9 (7.92)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.95 (3.069) | 24.51 (3.266) | 24.23 (3.173)

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity Screening Incidence to Detect the Presence of Anti-PegG-CSF Antibodies.
Description: Immunogenicity (anti-drug antibody; ADA) data is presented for all subjects' samples collected and a descriptive analysis is provided for immunogenicity (ADA) data.
  Percentage incidence within + 10% of the expected ADA positivity incidence of Test (6% ADA in Test is anticipated from literature) is not considered clinically significant.
  Evaluation of immunogenicity is carried out in a tiered fashion:
  1. Screening assay to assess if samples were positive or negative for anti-PegG-CSF.
  2. Confirmatory assays for samples that were positive in the screening assay. The confirmatory assays assessed if antibodies were specific for INTP5, Neulasta, PEG and/or filgrastim.
  3. Titer assay was performed to determine titer of the anti-PEG-GCSF antibody samples.
  4. Neutralizing antibody (NAb) assay for those samples that were positive in the confirmatory assays to assess the neutralizing capability of the antibody to inhibit pegfilgrastim activity.
Time Frame: Samples (8 mL each) were withdrawn at screening, at pre-dose and at 336 (D-15, Week 2), 504 (D-22, Week 3, within 60 minutes before 2nd dose), 840 (D-36, Week 5), 1176 (D-50, Week 7), 1680 (D-71, Week 10) and 2016 (D-85, Week 12) hours after first dose.
Measure: Count of Participants; unit: Participants
Arm/Group | INTP5 Biosimilar Product | US Neulasta Reference Product
Number analyzed (Participants) | 94 | 100
Participants
  Positive for Anti-Drug-Antibody | 10 | 9
  Positive in Neutralizing Anti-Drug-Antibody | 0 | 0
  No Anit-Drug Antibody Confirmed Positive Results | 84 | 91

2. Secondary Outcome: PK Endpoints: Pegfilgrastim C[Max]
Description: Pharmacokinetic (PK) properties of the test and reference formulations were assessed by measuring serum Pegfilgrastim concentration.
  Maximum measured serum concentration, calculated from the serum concentration vs. time profile of the individual subjects.
Time Frame: Venous blood samples (4 mL each) were withdrawn at pre-dose and at 8, 16, 24 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 120 (Day 6), 144 (Day 7), 240 (Day 11), 336 (Day 15) and 504 (Day 22) hours following 1st and 2nd dose, administration.
Population: All the 19 ADA confirmed positive subjects were included in the PK analysis: 10 subjects from INTP5 and 9 subjects from US-Neulasta.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- INTP5 Dose 1; INTP5 Dose 2: INTP5 subcutaneously at a dose of 6 mg/0.6 mL.
  INTP5: A pegfilgrastim biosimilar to US Neulasta.
- US Neulasta Dose 1; US Neulasta Dose 2: US Neulasta subcutaneously at a dose of 6 mg/0.6 mL.
  US Neulasta: FDA approved pegfilgrastim innovator product.
Arm/Group | INTP5 Dose 1 | INTP5 Dose 2 | US Neulasta Dose 1 | US Neulasta Dose 2
Number analyzed (Participants) | 10 | 10 | 9 | 9
ng/mL | 483.230 (175.1787) | 346.018 (150.4879) | 368.569 (223.3380) | 371.778 (263.4440)

3. Secondary Outcome: PK Endpoints: Pegfilgrastim AUC[0-t]
Description: Area under the serum concentration vs. time curve, calculated by linear trapezoidal rule from measured data points from the time zero to the time of last quantified concentration.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | INTP5 Dose 1 | INTP5 Dose 2 | US Neulasta Dose 1 | US Neulasta Dose 2
Number analyzed (Participants) | 10 | 10 | 9 | 9
ng.h/mL | 22417.938 (9922.2648) | 13640.695 (6709.2752) | 16610.870 (11255.1296) | 15255.327 (11050.7580)

4. Secondary Outcome: PK Endpoints: Pegfilgrastim AUC[0-∞]
Description: Area under the serum concentration versus time curve from time zero to infinity. Where AUC[0-infinity]= AUC[0-t] + Ct/lambda-z, Ct is the last measurable concentration and lamda-z is the terminal rate constant. AUC[0-infinity] is the sum of measurable and extrapolated parts.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | INTP5 Dose 1 | INTP5 Dose 2 | US Neulasta Dose 1 | US Neulasta Dose 2
Number analyzed (Participants) | 10 | 10 | 9 | 9
ng.h/mL | 22436.497 (9922.4383) | 13637.403 (6699.9736) | 16630.861 (11253.7406) | 15280.376 (11058.1142)

5. Secondary Outcome: PK Endpoints: Pegfilgrastim T[Max]
Description: The time of observing the peak concentration, calculated from the serum concentration vs. time profile of the individual subjects.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | INTP5 Dose 1 | INTP5 Dose 2 | US Neulasta Dose 1 | US Neulasta Dose 2
Number analyzed (Participants) | 10 | 10 | 9 | 9
h | 22.405 (3.3758) | 20.800 (5.5936) | 22.226 (3.5298) | 23.111 (2.6667)

6. Secondary Outcome: PK Endpoints: Pegfilgrastim λz (Lambda-z)
Description: Terminal rate constant: First order rate constant associated with the terminal (log-linear) portion of the curve. This was estimated via linear regression of time vs. log concentration. This parameter was calculated by linear least squares regression analysis using last three or more nonzero plasma concentration values.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | INTP5 Dose 1 | INTP5 Dose 2 | US Neulasta Dose 1 | US Neulasta Dose 2
Number analyzed (Participants) | 10 | 10 | 9 | 9
1/h | 0.021 (0.0071) | 0.025 (0.0142) | 0.022 (0.0058) | 0.019 (0.0074)

7. Secondary Outcome: PK Endpoints: Pegfilgrastim R^2 Adjusted
Description: Goodness of fit statistic for the terminal phase, adjusted for the number of points used in the estimation of λz (lambda-z). R^2 is the coefficient of determination and can range from 0 to 1, with higher values indicating greater predictability.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Coefficient of Determination
Arm/Group | INTP5 Dose 1 | INTP5 Dose 2 | US Neulasta Dose 1 | US Neulasta Dose 2
Number analyzed (Participants) | 10 | 10 | 9 | 9
Coefficient of Determination | 0.968 (0.0379) | 0.876 (0.133) | 0.974 (0.0245) | 0.879 (0.2339)

8. Secondary Outcome: PK Endpoints: Pegfilgrastim AUC[_%Extrap_Obs]
Description: The residual area in percentage determined by the formula, [(AUC[0-infinity]-AUC[0-t])/AUC[0-infinity]] x 100.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of AUC
Arm/Group | INTP5 Dose 1 | INTP5 Dose 2 | US Neulasta Dose 1 | US Neulasta Dose 2
Number analyzed (Participants) | 10 | 10 | 9 | 9
percentage of AUC | 0.115 (0.1106) | 0.644 (1.4428) | 0.230 (0.2672) | 0.266 (0.2664)

9. Secondary Outcome: PK Endpoints: Pegfilgrastim t[1/2]
Description: The terminal half-life calculated using the formula 0.693/(lambda-z)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | INTP5 Dose 1 | INTP5 Dose 2 | US Neulasta Dose 1 | US Neulasta Dose 2
Number analyzed (Participants) | 10 | 10 | 9 | 9
h | 36.721 (11.0052) | 36.612 (19.6215) | 34.172 (8.8669) | 40.616 (14.6054)

10. Secondary Outcome: PD Endpoints for Baseline Non-adjusted ANC: E[Max]
Description: Maximum measured absolute neutrophil count (ANC).
Time Frame: Venous blood samples (2 mL each) were withdrawn at pre-dose and at 8, 16, 24 (Day 2), 48 (Day 3), 72 (Day 4), 96 (Day 5), 120 (Day 6), 144 (Day 7), 240 (Day 11), 336 (Day 15) and 504 (Day 22) following 1st and 2nd dose administration.
Population: Outcome Measure Data Table is breaks participants into negative-ADA or positive-ADA, totaling the overall number of participants by arm
Measure: Mean (Standard Deviation); unit: x10^3cells/uL
Arm/Group | INTP5 Dose 1 | INTP5 Dose 2 | US Neulasta Dose 1 | US Neulasta Dose 2
Number analyzed (Participants) | 89 | 89 | 93 | 93
x10^3cells/uL
  ADA-NEGATIVE: number analyzed (Participants) | 79 | 79 | 84 | 84
  ADA-NEGATIVE | 40.72 (10.862) | 44.63 (11.077) | 38.34 (9.925) | 40.62 (8.963)
  ADA-POSITIVE: number analyzed (Participants) | 10 | 10 | 9 | 9
  ADA-POSITIVE | 42.89 (10.512) | 46.53 (9.093) | 38.38 (8.211) | 44.96 (16.409)

11. Secondary Outcome: PD Endpoints for Baseline Non-adjusted ANC: T[Max]
Description: Area under the ANC versus time curve from time zero to the last measurable concentration as calculated by linear trapezoidal method.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: h
Arm/Group | INTP5 Dose 1 | INTP5 Dose 2 | US Neulasta Dose 1 | US Neulasta Dose 2
Number analyzed (Participants) | 89 | 89 | 93 | 93
h
  ADA-NEGATIVE: number analyzed (Participants) | 79 | 79 | 84 | 84
  ADA-NEGATIVE | 64.710 (11.1076) | 59.587 (14.9170) | 63.182 (15.8763) | 64.637 (20.5772)
  ADA-POSITIVE: number analyzed (Participants) | 10 | 10 | 9 | 9
  ADA-POSITIVE | 72.003 (0.0072) | 67.453 (15.7091) | 64.002 (12.0014) | 61.461 (29.9401)

12. Secondary Outcome: PD Endpoints for Baseline Non-adjusted ANC: AUEC[0-t]
Description: Time to reach the maximum measured absolute neutrophil count (ANC)
Time Frame: as for outcome 10
Population: Table breaks participants into ADA(-) or ADA(+), totaling the overall number of participants by arm. 5 Subjects having three consecutive missing samples in elimination phase were excluded from the analysis of AUEC0-t reducing the total participants to 88 for INTP5 Dose 1, 88 for INTP5 Dose 2, 92 for Neulasta Dose 1, and 91 for Neulasta Dose 2.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | INTP5 Dose 1 | INTP5 Dose 2 | US Neulasta Dose 1 | US Neulasta Dose 2
Number analyzed (Participants) | 88 | 88 | 92 | 91
h*ng/mL
  ADA-NEGATIVE: number analyzed (Participants) | 78 | 79 | 83 | 82
  ADA-NEGATIVE | 7107.14 (1481.971) | 7929.25 (1561.246) | 6718.70 (1361.957) | 7359.09 (1455.570)
  ADA-POSITIVE: number analyzed (Participants) | 10 | 9 | 9 | 9
  ADA-POSITIVE | 7286.53 (1744.737) | 8539.99 (1522.935) | 6846.77 (763.675) | 7761.65 (1658.478)

13. Secondary Outcome: PD Endpoints for Baseline Adjusted ANC: E[Max]
Description: Maximum measured absolute neutrophil count (ANC).
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: x10^3cells/uL
Arm/Group | INTP5 Dose 1 | INTP5 Dose 2 | US Neulasta Dose 1 | US Neulasta Dose 2
Number analyzed (Participants) | 88 | 88 | 91 | 89
x10^3cells/uL
  ADA-NEGATIVE: number analyzed (Participants) | 78 | 78 | 82 | 80
  ADA-NEGATIVE | 36.50 (10.458) | 40.80 (11.038) | 33.35 (9.189) | 36.56 (8.755)
  ADA-POSITIVE: number analyzed (Participants) | 10 | 10 | 9 | 9
  ADA-POSITIVE | 38.37 (9.548) | 42.50 (10.061) | 34.18 (8.503) | 40.76 (17.170)

14. Secondary Outcome: PD Endpoints for Baseline Adjusted ANC: AUEC[0-t]
Description: Area under the absolute neutrophil count (ANC) versus time curve from time zero to the last measurable concentration as calculated by linear trapezoidal method.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: x10^3cells*h/uL
Arm/Group | INTP5 Dose 1 | INTP5 Dose 2 | US Neulasta Dose 1 | US Neulasta Dose 2
Number analyzed (Participants) | 87 | 87 | 90 | 89
x10^3cells*h/uL
  ADA-NEGATIVE: number analyzed (Participants) | 77 | 78 | 81 | 80
  ADA-NEGATIVE | 4920.26 (1339.674) | 5992.49 (1555.062) | 4389.55 (1140.655) | 5441.01 (1478.241)
  ADA-POSITIVE: number analyzed (Participants) | 10 | 9 | 9 | 9
  ADA-POSITIVE | 4967.86 (1229.792) | 6539.58 (2202.473) | 4578.32 (1200.125) | 5676.92 (1991.456)

15. Secondary Outcome: PD Endpoints for Baseline Adjusted ANC: T[Max]
Description: Time to reach the maximum measured absolute neutrophil count (ANC)
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: h
Arm/Group | INTP5 Dose 1 | INTP5 Dose 2 | US Neulasta Dose 1 | US Neulasta Dose 2
Number analyzed (Participants) | 88 | 88 | 91 | 91
h
  ADA-NEGATIVE: number analyzed (Participants) | 78 | 78 | 82 | 82
  ADA-NEGATIVE | 64.617 (11.1482) | 59.735 (14.9546) | 65.553 (15.8887) | 65.043 (20.6610)
  ADA-POSITIVE: number analyzed (Participants) | 10 | 10 | 9 | 9
  ADA-POSITIVE | 72.003 (0.0072) | 67.453 (15.7091) | 64.002 (12.0014) | 61.461 (29.9401)

16. Secondary Outcome: PD Endpoints for Baseline Adjusted ANC: λz (Lambda-z)
Description: First order rate constant associated with the terminal (log-linear) portion of the curve. This was estimated via linear regression of time vs. log concentration. This parameter was calculated by linear least squares regression analysis using last three or more non-zero plasma concentration values.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: h
Arm/Group | INTP5 Dose 1 | INTP5 Dose 2 | US Neulasta Dose 1 | US Neulasta Dose 2
Number analyzed (Participants) | 86 | 87 | 89 | 88
h
  ADA-NEGATIVE: number analyzed (Participants) | 76 | 78 | 80 | 79
  ADA-NEGATIVE | 0.01 (0.007) | 0.01 (0.006) | 0.01 (0.006) | 0.01 (0.006)
  ADA-POSITIVE: number analyzed (Participants) | 10 | 9 | 9 | 9
  ADA-POSITIVE | 0.01 (0.006) | 0.01 (0.003) | 0.01 (0.004) | 0.01 (0.005)

17. Secondary Outcome: PD Endpoints for Baseline Adjusted ANC: t[1/2]
Description: The terminal half-life will be calculated as 0.693/(lambda-z)
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: h
Arm/Group | INTP5 Dose 1 | INTP5 Dose 2 | US Neulasta Dose 1 | US Neulasta Dose 2
Number analyzed (Participants) | 86 | 87 | 89 | 88
h
  ADA-NEGATIVE: number analyzed (Participants) | 76 | 78 | 80 | 79
  ADA-NEGATIVE | 62.25 (28.847) | 64.13 (26.785) | 77.23 (86.239) | 76.02 (59.888)
  ADA-POSITIVE: number analyzed (Participants) | 10 | 9 | 9 | 9
  ADA-POSITIVE | 67.03 (41.296) | 69.72 (25.447) | 81.74 (29.981) | 67.02 (22.706)

ADVERSE EVENTS:
Time Frame: 99 Days
Arm/Group | INTP5 Biosimilar Product | US Neulasta Reference Product
All-Cause Mortality (participants affected / at risk) | 0/100 | 1/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 1/100
Other Adverse Events (participants affected / at risk) | 32/100 | 37/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INTP5 Biosimilar Product (N=100) | US Neulasta Reference Product (N=100)
death (General disorders) | 0 (0) | 1 (1) — There was 1 death reported. The subject died due to accidental drowning. The AE was severe in nature and the relationship of the AE to the study drug was considered as not related. Apart from the death, no other SAEs were reported during the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INTP5 Biosimilar Product (N=100) | US Neulasta Reference Product (N=100)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (7) | 5 (7)
Chills (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 5 (5) | 4 (4)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Eosinophil count increased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Human chorionic gonadotropin increased (Investigations) | 0 (0) | 1 (1)
Protein urine present (Investigations) | 1 (1) | 1 (1)
Red blood cells urine positive (Investigations) | 3 (3) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 16 (17) | 15 (16)
Headache (Nervous system disorders) | 6 (7) | 13 (13)
Urine abnormality (Investigations) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT04015232/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/32/NCT04015232/SAP_001.pdf